CLINICAL TRIAL: NCT04948528
Title: Diagnostic Evaluation of Urine DNA Methylation/Somatic Mutation Profiling for Upper Tract Urothelial Carcinoma Detection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AnchorDx Medical Co., Ltd. (Industry)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Peking University First Hospital (Other); Peking University Third Hospital (Other); Peking Union Medical College Hospital (Other); The Affiliated Hospital of Qingdao University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Sir Run Run Shaw Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Other Study IDs: AnchorDx BC006
Record Dates: First submitted 2021-06-22; First posted 2021-07-02 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Upper Tract Urothelial Carcinoma
Keywords: upper tract urothelial carcinoma; urine; DNA methylation; somatic mutation
MeSH Terms: interventions — Cystoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — First void and non-first-void urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group:: All suspected upper tract urothelial carcinoma participants will be assigned to case group.
  Interventions: Other: Active Comparator: Surgery Pathology or Cystoscopy
- Control group: All suspected upper tract urothelial benign participants such as ureteral/renal calculi, ureteral stricture, upper urinary tract polyps, pyelonephritis, urinary tuberculosis will be assigned to control group.
  Interventions: Other: Active Comparator: Clinical Diagnosis

INTERVENTIONS:
Other: Active Comparator: Surgery Pathology or Cystoscopy — Case group will be followed up with surgery pathology or cystoscopy.
  Groups: Case group:
Other: Active Comparator: Clinical Diagnosis — Control group will be diagnosed in clinical.
  Groups: Control group

SUMMARY:
Clinical trial to determine the efficacy (sensitivity and specificity) of Anchordx's urine DNA methylation/somatic mutation assay for detecting upper tract urothelial carcinoma compared to pathology in patients.

DETAILED DESCRIPTION:
This is a prospective study that involves 8 centers in China and 490 participants. The test analyzes the DNA methylation/somatic mutation profiles of urothelial cancer-specific biomarkers non-invasively using urine specimens collected before invasive diagnosis/treatment. The efficacy (sensitivity and specificity) of the assay for detection of upper tract urothelial carcinoma is evaluated in comparison to pathology or cystoscopy.

ELIGIBILITY:
Inclusion Criteria:

Case group:

* 1.Any male or female patient aged 18 or older.
* 2.Able to provide urine specimen (100ml for both first void and non-first-void urine) before treatments.
* 3.Diagnosed with incident upper tract urothelial carcinoma (including renal pelvis carcinoma and ureteral carcinoma) by surgery.
* 4.Able to provide legally effective informed consent.

Control group:

* 1.Any male or female patient aged 18 or older.
* 2.Able to provide urine specimen (100ml for both first void and non-first-void urine) before treatments.
* 3.Diagnosed with urinary disease such as ureteral/renal calculi, ureteral stricture, upper urinary tract polyps, pyelonephritis, urinary tuberculosis.
* 4.Able to provide legally effective informed consent.

Exclusion Criteria:

* 1.Patients had been diagnosed with cancer history.
* 2.Patients diagnosed with cancers unmatched with inclusion criteria cancers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: suspected upper tract urothelial carcinoma patients
Sampling Method: Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-06-25 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of urine DNA methylation/somatic mutation test | 1 Year
  Sensitivity and specificity of urine DNA methylation/somatic mutation test (the proportion of pathology that are correctly identified as such by pathology)

CONTACTS AND LOCATIONS:
Overall Officials: Jian HUANG, MD, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No